CLINICAL TRIAL: NCT00781586
Title: A Randomized, Single Center, Double-blind, Three-way Crossover Trial to Evaluate the Efficacy of ONE A DAY Weightsmart Advanced Versus Caffeine and Placebo on Energy Expenditure, Thermogenesis and Perceived Energy Levels in Women.
Brief Title: Efficacy of ONE A DAY Weightsmart Advanced Versus Caffeine and Placebo on Energy Expenditure, Thermogenesis and Perceived Energy Levels in Women.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 12956
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Energy Expenditure
Keywords: Energy expenditure; Nutritional; Weight control
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Dietary Supplement: One-A-Day Weight S.A. (Multi-Vitamins, BAY94-9350)
- Arm 2 (Active Comparator)
  Interventions: Drug: Caffeine
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: One-A-Day Weight S.A. (Multi-Vitamins, BAY94-9350) — One A Day Weight Smart Advanced 1 tablet at 1st visit
  Arms: Arm 1
Drug: Caffeine — Caffeine 100 mg 1 tablet at 1st visit
  Arms: Arm 2
Drug: Placebo — Placebo 1 tablet at 1st visit
  Arms: Arm 3

SUMMARY:
The study is considered research because efficacy (how well a drug works) information is needed in healthy, 25-45 year-old, female subjects with moderate caffeine intake. The investigational product is available in the United States without a prescription (over-the-counter) as a nutritional supplement. The purpose of this study is to assess whether One-A-Day Weightsmart Advanced is safe and can increase metabolism and perceived energy in female subjects compared with caffeine or placebo (inactive drug). Participation in this study will last approximately 4 weeks and require about 4 outpatient visits to St. Luk's-Roosevelt Hospital Center. About 21 subjects are expected to participate in this study.

DETAILED DESCRIPTION:
- Primary efficacy endpoints are area under the curve (AUC) over the first 2 hours and the last 2 hours of Resting Metabolic RateRespiratory Quotient- The secondary efficacy endpoints are:Perceived Energy scales Visual Analog Scale (VAS) Change from baseline for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) respiration, average heart rate over 1st 20 minutes, average heart rate over last 20 minutes, and temperature

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy, ambulatory female between the ages of 25 and 45 years old with a Body Mass Index (BMI) between 20 and 35 kg/m2 (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, brief physical examination, including vital signs, and clinical laboratory tests)
* Consume a habitual caffeine intake (<300 mg/day or </= 2 caffeinated drinks/day)

Exclusion Criteria:

* Pregnant, planning to become pregnant or lactating females
* Using ephedra- or caffeine-containing products or chronic medications other than contraceptives or HRT
* Lost or gained more than five pounds of weight in the preceding three months
* Engage in intense physical activities
* Use of tobacco or nicotine products
* A medical history with known thyroid disease, blood pressure >140/90 mmHg, diabetes, depression, psychiatric disorders, glaucoma, or seizure disorders and other relevant illnesses that can interfere with the trial in the opinion of the Investigator

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-10-02 (Actual); Primary Completion 2008-04-21 (Actual); Study Completion 2008-04-21 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of RMR for the first 2 hours | Primary efficacy endpoints are area under the curve (AUC) over the first 2 hours and the last 2 hours of Resting Metabolic Rate and Respiratory Quotient
AUC of RMR for the last 2 hours | Primary efficacy endpoints are area under the curve (AUC) over the first 2 hours and the last 2 hours of Resting Metabolic Rate and Respiratory Quotient
AUC of Respiratory Quotient (RQ) for the first 2 hours | Primary efficacy endpoints are area under the curve (AUC) over the first 2 hours and the last 2 hours of Resting Metabolic Rate and Respiratory Quotient
AUC of RQ for the last 2 hours | Primary efficacy endpoints are area under the curve (AUC) over the first 2 hours and the last 2 hours of Resting Metabolic Rate and Respiratory Quotient

SECONDARY OUTCOMES:
Perceived Energy scales - Visual Analog Scale (VAS) | Change from baseline for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) respiration, average heart rate over 1st 20 minutes, average heart rate over last 20 minutes, and temperature
AUC for heart rate for the first 2 hours | Change from baseline for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) respiration, average heart rate over 1st 20 minutes, average heart rate over last 20 minutes, and temperature
AUC for heart rate for the last 2 hours | Change from baseline for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) respiration, average heart rate over 1st 20 minutes, average heart rate over last 20 minutes, and temperature
Change from baseline for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), respiration and temperature | Change from baseline for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) respiration, average heart rate over 1st 20 minutes, average heart rate over last 20 minutes, and temperature

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- New York, New York, United States